CLINICAL TRIAL: NCT02348216
Title: A Phase 1/2 Multicenter Study Evaluating the Safety and Efficacy of KTE-C19 in Adults With Refractory Aggressive Non-Hodgkin Lymphoma
Brief Title: Study Evaluating the Safety and Efficacy of KTE-C19 in Adult Participants With Refractory Aggressive Non-Hodgkin Lymphoma
Acronym: ZUMA-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KTE-C19-101; 2015-005007-86 (EudraCT Number)
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Results first posted 2021-11-23 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Refractory Diffuse Large B Cell Lymphoma (DLBCL); Relapsed Diffuse Large B-Cell Lymphoma; Transformed Follicular Lymphoma (TFL); Primary Mediastinal B-cell Lymphoma (PMBCL); High Grade B-cell Lymphoma (HGBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — axicabtagene ciloleucel; fludarabine; Cyclophosphamide; Levetiracetam; tocilizumab; Dexamethasone; Methylprednisolone; Bendamustine Hydrochloride; Rituximab; Doxorubicin; Prednisone; Vincristine; Ifosfamide; Carboplatin; Etoposide; Gemcitabine; Oxaliplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 1 Study: Axicabtagene Ciloleucel and Conditioning Chemotherapy (Experimental): Participants with diffuse large B-cell lymphoma (DLBCL), primary mediastinal B-cell lymphoma (PMBCL), or transformed follicular lymphoma (TFL) will receive conditioning chemotherapy (fludarabine 30 mg/m^2 intravenously [IV] over 30 minutes and cyclophosphamide 500 mg/m^2 IV over 60 minutes) on Days -5, -4, and -3; followed by a single infusion of axicabtagene ciloleucel chimeric antigen receptor (CAR) transduced autologous T cells administered IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of body weight (BW) on Day 0.
  Interventions: Biological: Axicabtagene Ciloleucel; Drug: Fludarabine; Drug: Cyclophosphamide
- Phase 2 (Pivotal Study): Cohort 1 (Experimental): Participants with refractory DLBCL will receive conditioning chemotherapy (fludarabine 30 mg/m^2 IV over 30 minutes and cyclophosphamide 500 mg/m^2 IV over 60 minutes) on Days -5, -4, and -3; followed by a single infusion of axicabtagene ciloleucel CAR transduced autologous T cells administered IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of BW on Day 0.
  Interventions: Biological: Axicabtagene Ciloleucel; Drug: Fludarabine; Drug: Cyclophosphamide
- Phase 2 (Pivotal Study): Cohort 2 (Experimental): Participants with refractory PMBCL or TFL will receive conditioning chemotherapy (fludarabine 30 mg/m^2 IV over 30 minutes and cyclophosphamide 500 mg/m^2 IV over 60 minutes) on Days -5, -4, and -3; followed by a single infusion of axicabtagene ciloleucel CAR transduced autologous T cells administered IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of BW on Day 0.
  Interventions: Biological: Axicabtagene Ciloleucel; Drug: Fludarabine; Drug: Cyclophosphamide
- Phase 2 (Safety Management Study): Cohort 3 (Experimental): Participants with relapsed or refractory transplant ineligible DLBCL, PMBCL, or TFL will receive conditioning chemotherapy (fludarabine 30 mg/m^2 IV over 30 minutes and cyclophosphamide 500 mg/m^2 IV over 60 minutes) on Days -5, -4, and -3; followed by a single infusion of axicabtagene ciloleucel CAR transduced autologous T cells administered IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of BW on Day 0. Participants will also receive a prophylactic regimen of levetiracetam (750 mg orally or IV twice daily (BID) starting on Day 0) and tocilizumab (8 mg/kg IV over 1 hour (not to exceed 800 mg)) on Day 2).
  Interventions: Biological: Axicabtagene Ciloleucel; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Levetiracetam; Drug: Tocilizumab
- Phase 2 (Safety Management Study): Cohort 4 (Experimental): Participants with r/r DLBCL,PMBCL,TFL,or high-grade B-cell lymphoma(HGBCL)after 2 systemic lines of therapy will receive optional bridging therapy(dexamethasone 20mg to 40mg,eitherorally or IV daily for 1 to 4 days or 1g/m^2 of high-dose methylprednisolone(HDMP)for 3 days with rituximab at 375mg/m^2 weekly for 3 weeks or bendamustine 90 mg/m^2 on Days 1 and 2 and rituximab 375mg/m^2 on Day 1),conditioning chemotherapy(fludarabine 30mg/m^2 IV and cyclophosphamide 500mg/m^2 IV)on Days -5,-4, and -3;followed by single infusion of axicabtagene ciloleucel CAR transduced autologous T cells IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of BW. Participants will receive a prophylactic regimen of levetiracetam(750 mg orally or IV twice daily(BID)starting on Day 0).Participants will receive tocilizumab(initiated on persistent Grade 1 cytokine release syndrome(CRS)for over 24 hours)and dexamethasone(persistent Grade 1 CRS for over 72 hours and at onset of Grade 1 neurologic toxicity).
  Interventions: Biological: Axicabtagene Ciloleucel; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Levetiracetam; Drug: Tocilizumab; Drug: Dexamethasone; Drug: High-dose methylprednisolone; Drug: Bendamustine; Drug: Rituximab
- Phase 2 (Safety Management Study): Cohort 5 (Experimental): Participants with r/r DLBCL, PMBCL ,TFL, or HGBCL after 2 systemic lines of therapy will receive debulking therapy (R-CHOP:rituximab 375mg/m^2 D1,doxorubicin 50mg/m^2 D1,prednisone 100mg D1 to D5,cyclophosphamide 750mg/m^2 D1,vincristine 1.4 mg/m^2 D1 or R-ICE:rituximab 375mg/ m^2 D1,ifosfamide 5g/m^2 24h-CI D2,carboplatin AUC5 D2 maximum dose 800mg,etoposide 100 mg/m^2/day D1 to D3 or R-GEMOX:rituximab 375mg/m^2 D1,gemcitabine 1000mg/m^2 D2,oxaliplatin 100mg/m^2 D2 or R-GDP:rituximab 375mg/m^2 D1 or D8,gemcitabine 1g/m^2 D1 & D8,dexamethasone 40mg D1 to D4,cisplatin 75mg/m^2 D1(or carboplatin AUC5 D1) or radiotherapy:20 to 30 Gy), conditioning chemotherapy (fludarabine 30mg/m^2 IV and cyclophosphamide 500mg/m^2 IV)on Days -5,-4, and -3; followed by single infusion of axicabtagene ciloleucel at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of BW on Day 0. Participants will also receive a prophylactic regimen of levetiracetam (750 mg orally or IV BID starting on D0).D=Day.
  Interventions: Biological: Axicabtagene Ciloleucel; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Levetiracetam; Drug: Rituximab; Drug: Doxorubicin; Drug: Prednisone; Drug: Vincristine; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Cisplatin
- Phase 2 (Safety Management Study): Cohort 6 (Experimental): Participants with r/r DLBCL,PMBCL,TFL orHGBCL after 2 systemic lines of therapy may receive bridging therapy(dexamethasone 20mg to 40mg,orally or IV daily for 1 to 4 days or 1g/m^2 HDMP for 3 days with rituximab at 375mg/m^2 weekly for 3 weeks or bendamustine 90 mg/m^2 on Days 1 and 2 and rituximab 375mg/m^2 on Day 1),conditioning chemotherapy(fludarabine 30mg/m^2 IV and cyclophosphamide 500mg/m^2 IV)on Days -5,-4, and -3; followed by single infusion of axicabtagene ciloleucel CAR transduced autologous T cells IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of BW on Day 0.Participants will also receive a prophylactic regimen of levetiracetam 750 mg orally or IV twice daily(BID)starting on Day 0)and corticosteroids(dexamethasone, 10 mg once daily on Days 0, 1, and 2).Participants will receive tocilizumab(initiated on persistent Grade 1 CRS for over 24 hours)and dexamethasone(persistent Grade 1 CRS for over 72 hours and at onset of Grade 1 neurologic toxicity).
  Interventions: Biological: Axicabtagene Ciloleucel; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Levetiracetam; Drug: Tocilizumab; Drug: Dexamethasone; Drug: High-dose methylprednisolone; Drug: Bendamustine; Drug: Rituximab; Drug: Methylprednisolone

INTERVENTIONS:
Biological: Axicabtagene Ciloleucel — A single infusion of chimeric antigen receptor (CAR)-transduced autologous T cells administered intravenously at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg.
  Other Names: Yescarta®
Drug: Fludarabine — Administered according to package insert
Drug: Cyclophosphamide — Administered according to package insert
Drug: Levetiracetam — Administered according to package insert
  Arms: Phase 2 (Safety Management Study): Cohort 3; Phase 2 (Safety Management Study): Cohort 4; Phase 2 (Safety Management Study): Cohort 5; Phase 2 (Safety Management Study): Cohort 6
Drug: Tocilizumab — Administered according to package insert
  Arms: Phase 2 (Safety Management Study): Cohort 3; Phase 2 (Safety Management Study): Cohort 4; Phase 2 (Safety Management Study): Cohort 6
Drug: Dexamethasone — Administered according to package insert
  Arms: Phase 2 (Safety Management Study): Cohort 4; Phase 2 (Safety Management Study): Cohort 6
Drug: High-dose methylprednisolone — Administered according to package insert
  Arms: Phase 2 (Safety Management Study): Cohort 4; Phase 2 (Safety Management Study): Cohort 6
Drug: Bendamustine — Administered according to package insert
  Arms: Phase 2 (Safety Management Study): Cohort 4; Phase 2 (Safety Management Study): Cohort 6
Drug: Rituximab — Administered according to package insert
  Arms: Phase 2 (Safety Management Study): Cohort 4; Phase 2 (Safety Management Study): Cohort 5; Phase 2 (Safety Management Study): Cohort 6
Drug: Doxorubicin — Administered according to package insert
  Arms: Phase 2 (Safety Management Study): Cohort 5
Drug: Prednisone — Administered according to package insert
  Arms: Phase 2 (Safety Management Study): Cohort 5
Drug: Vincristine — Administered according to package insert
  Arms: Phase 2 (Safety Management Study): Cohort 5
Drug: Ifosfamide — Administered according to package insert
  Arms: Phase 2 (Safety Management Study): Cohort 5
Drug: Carboplatin — Administered according to package insert
  Arms: Phase 2 (Safety Management Study): Cohort 5
Drug: Etoposide — Administered according to package insert
  Arms: Phase 2 (Safety Management Study): Cohort 5
Drug: Gemcitabine — Administered according to package insert
  Arms: Phase 2 (Safety Management Study): Cohort 5
Drug: Oxaliplatin — Administered according to package insert
  Arms: Phase 2 (Safety Management Study): Cohort 5
Drug: Cisplatin — Administered according to package insert
  Arms: Phase 2 (Safety Management Study): Cohort 5
Drug: Methylprednisolone — Administered according to package insert
  Arms: Phase 2 (Safety Management Study): Cohort 6

SUMMARY:
This study will be separated into 3 distinct phases designated as the Phase 1 study, Phase 2 pivotal study (Cohort 1 and Cohort 2), and Phase 2 safety management study (Cohort 3 and Cohort 4, Cohort 5 and Cohort 6).

The primary objectives of this study are:

* Phase 1 Study: Evaluate the safety of axicabtagene ciloleucel regimens
* Phase 2 Pivotal Study; Evaluate the efficacy of axicabtagene ciloleucel
* Phase 2 Safety Management Study: Assess the impact of prophylactic regimens or earlier interventions on the rate and severity of cytokine release syndrome (CRS) and neurologic toxicities

Subjects who received an infusion of KTE-C19 will complete the remainder of the 15 year follow-up assessments in a separate long-term follow-up study, KT-US-982-5968.

ELIGIBILITY:
Key Inclusion Criteria

1. Histologically confirmed:

   * Diffuse Large B Cell Lymphoma (DLBCL)
   * Primary Mediastinal Large B Cell Lymphoma (PMBCL)
   * Transformation Follicular Lymphoma (TFL)
   * High grade B-cell lymphoma (HGBCL)
2. Chemotherapy-refractory disease, defined as one of more of the following:

   * No response to last line of therapy i. Progressive disease (PD) as best response to most recent therapy regimen ii. Stable disease (SD) as best response to most recent therapy with duration no longer than 6 month from last dose of therapy OR
   * Refractory post-autologous stem cell transplant (ASCT) i. Disease progression or relapsed less than or equal to 12 months of ASCT (must have biopsy proven recurrence in relapsed individuals) ii. If salvage therapy is given post-ASCT, the individual must have had no response to or relapsed after the last line of therapy
3. Individuals must have received adequate prior therapy including at a minimum:

   * Anti-cluster of differentiate 20 (CD20) monoclonal antibody unless investigator determines that tumor is CD20-negative and
   * an anthracycline containing chemotherapy regimen
   * for individual with transformed FL must have chemorefractory disease after transformation to DLBCL.
4. At least one measurable lesion per revised international working group (IWG Response Criteria
5. Eastern cooperative oncology group (ECOG) performance status of 0 or 1
6. Absolute neutrophil count (ANC) ≥ 1000/microliters (uL)
7. Absolute lymphocyte count ≥ 100/uL
8. Platelet count ≥ 75,000/uL
9. Adequate renal, hepatic, pulmonary and cardiac function defined as:

   * Creatinine clearance (as estimated by Cockcroft Gault) > 60 mL/min
   * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) < 2.5 upper limit of normal (ULN)
   * Total bilirubin < 1.5 mg/dL, except in individuals with Gilbert's syndrome
   * Cardiac ejection fraction >50%, no evidence of pericardial effusion as determined by an echocardiogram (ECHO), and no clinically significant pleural effusion
   * Baseline oxygen saturation >92% on room air
10. All individuals or legally appointed representatives/caregivers, must personally sign and date the Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved consent form before initiating any study specific procedures or activities.
11. Relapsed or refractory large B-cell lymphoma including DLBCL, PMBCL, TFL, and HGBCL after two systemic lines of therapy

Key Exclusion Criteria

1. History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) or follicular lymphoma unless disease free for at least 3 years
2. History of allogeneic stem cell transplantation
3. Prior chimeric antigen receptor (CAR) therapy or other genetically modified T cell therapy
4. Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous (IV) antimicrobials for management. Simple urinary tract infection (UTI) and uncomplicated bacterial pharyngitis are permitted if responding to active treatment
5. History of human immunodeficiency virus (HIV) infection or acute or chronic active hepatitis B or C infection. Individuals with history of hepatitis infection must have cleared their infection as determined by standard serological and genetic testing per current Infectious Diseases Society of America (IDSA) guidelines
6. Individuals with detectable cerebrospinal fluid malignant cells, or brain metastases, or with a history of central nervous system (CNS) lymphoma or primary CNS lymphoma, cerebrospinal fluid malignant cells or brain metastases
7. History or presence of CNS disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2015-04-21 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (36):
- United States (23):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope, Duarte, California
  - University of California San Diego (UCSD), La Jolla, California
  - Stanford University, Palo Alto, California
  - University of California Los Angeles (UCLA), Santa Monica, California
  - Sarah Cannon - Denver, Denver, Colorado
  - University of Miami, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - Sarah Cannon - Tennesee, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Sarah Cannon-Methodist Healthcare System - San Antonio, San Antonio, Texas
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Princess Margaret, Toronto, Ontario
- France (3):
  - Hopital Saint Louis, Paris
  - Hopital Haut-Leveque, Pessac
  - CHU de Rennes, Rennes
- Germany (3):
  - Universitätsklinik Dresden, Dresden
  - University Hospital of Essen, Essen
  - Universitaetsklinikum Wuerzburg, Würzburg
- Tel Aviv Souraski Medical Center, Tel Aviv, Israel
- Netherlands (4):
  - Academisch Medisch Centrum, Amsterdam
  - University Medical Center Groningen, Groningen
  - Erasmus MC, Rotterdam
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and transparency
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Topp MS, van Meerten T, Wermke M et al. Preliminary Results of Earlier Steroid Use with Axicabtagene Ciloleucel in Patients With Relapsed/Refractory Large B Cell Lymphoma. Poster presented at the American Society of Presented at: American Society of Clinical Oncology Annual Meeting. May 31-June 4, 2019; Chicago, Illinois; Abstract 7558.
- [Result] Topp, M, van Meerten T, Houot R, et al. (2019). Earlier Steroid Use with Axicabtagene Ciloleucel (Axi-Cel) in Patients with Relapsed/Refractory Large B Cell Lymphoma. Blood (ASH Annual Meeting Abstracts) 134(Suppl 1): 243. Abstract 626.
- [Result] Abstract: Oluwole OO, et al. Prophylactic corticosteroid use with axicabtagene ciloleucel in patients with relapsed/refractory large B-cell lymphoma. Transplantation and Cellular Therapy 2021.
- [Result] Oluwole OO, Bouabdallah K, Munoz J, De Guibert S, Vose JM, Bartlett NL, Lin Y, Deol A, McSweeney PA, Goy AH, Kersten MJ, Jacobson CA, Farooq U, Minnema MC, Thieblemont C, Timmerman JM, Stiff P, Avivi I, Tzachanis D, Kim JJ, Bashir Z, McLeroy J, Zheng Y, Rossi JM, Johnson L, Goyal L, van Meerten T. Prophylactic corticosteroid use in patients receiving axicabtagene ciloleucel for large B-cell lymphoma. Br J Haematol. 2021 Aug;194(4):690-700. doi: 10.1111/bjh.17527. Epub 2021 Jul 22. PMID 34296427
- [Result] Santa Monica, Calif. New Four-Year Data Show Long-Term Survival in Patients With Large B-Cell Lymphoma Treated With Yescarta® in ZUMA-1 Trial. Data presented at the 62nd American Society of Hematology (ASH) Annual Meeting and Exposition. December 5, 2020; Abstract 1187
- [Result] Max S. Topp, Tom van Meerten, Martin Wermke, Pieternella J. Lugtenburg, Monique C. Minnema, Kevin W. Song, Catherine Thieblemont, Yizhou Jiang, Vicki Plaks, Anne Kerber, Marie José Kersten. Preliminary Results of Earlier Steroid Use With Axicabtagene Ciloleucel in Patients With Relapsed/ Refractory Large B Cell Lymphoma. Poster presented at ASCO 2019 Annual Meeting. June 3, 2019; Abstract 7558
- [Result] Sattva S. Neelapu, Caron A. Jacobson, Olalekan O. Oluwole, Javier Munoz, Abhinav Deol, David B. Miklos, Nancy L. Bartlett, Ira Braunschweig, Yizhou Jiang, Jenny J. Kim, Lianqing Zheng, John M. Rossi, Frederick L. Locke. Axicabtagene Ciloleucel (Axi-Cel) In Refractory Large B Cell Lymphoma: Outcomes in Patients ≥ or < 65 Years of Age in the Pivotal Phase 1/2 ZUMA-1 Study. Poster presented at EHA 2019. June 15, 2019; Abstract 1066
- [Result] Max S. Topp, Tom van Meerten, Martin Wermke, Pieternella J. Lugtenburg, Monique C. Minnema, Kevin W. Song, Catherine Thieblemont, Yizhou Jiang, Vicki Plaks, Anne Kerber, Marie José Kersten. Axicabtagene Ciloleucel (Axi-Cel) in Patients With Relapsed/Refractory Large B Cell Lymphoma: Preliminary Results of Earlier Steroid Use. Poster presented at EHA 2019. June 15, 2019; Abstract 1067
- [Result] Sattva S. Neelapu, John M. Rossi, Caron A. Jacobson, Frederick L. Locke, David B. Miklos, Patrick M. Reagan, Scott Rodig, Lazaros J. Lekakis, Ian W. Flinn, Lianqing Zheng, Francesca Milletti, Edmund Chang, Allen Xue, Vicki Plaks, Jenny J. Kim, Adrian Bot. CD19-Loss With Preservation of Other B Cell Lineage Features in Patients With Large B Cell Lymphoma Who Relapsed Post-Axi-Cel. Blood (ASH Annual Meeting Abstracts) 134(Suppl 1): 203. Abstract 704.
- [Result] Sattva S. Neelapu, Frederick L. Locke, Nancy L. Bartlett, Lazaros J. Lekakis, Patrick Reagan, David B. Miklos, Caron A. Jacobson, Ira Braunschweig, Olalekan Oluwole, Tanya Siddiqi, Yi Lin, Michael Crump, John Kuruvilla, Eric Van Den Neste, Umar Farooq, Lynn Navale, Venita DePuy, Jenny J. Kim, Christian Gisselbrecht. A Comparison of Two-Year Outcomes in ZUMA-1 (Axicabtagene Ciloleucel) and SCHOLAR-1 in Patients With Refractory Large B Cell Lymphoma. Blood (ASH Annual Meeting Abstracts) 134(Suppl 1): 4095. Abstract 626.
- [Derived] Chartier M, Filosto S, Peyret T, Chiney M, Milletti F, Budka J, Ndi A, Dong J, Vardhanabhuti S, Mao D, Duffull S, Dodds M, Shen R. Investigating the Influence of Covariates on Axicabtagene Ciloleucel (axi-cel) Kinetics in Patients with Non-Hodgkin's Lymphoma. Clin Pharmacokinet. 2024 Sep;63(9):1283-1299. doi: 10.1007/s40262-024-01413-z. Epub 2024 Sep 6. PMID 39240498
- [Derived] Locke FL, Siddiqi T, Jacobson CA, Ghobadi A, Ahmed S, Miklos DB, Perales MA, Munoz J, Fingrut WB, Pennisi M, Gauthier J, Shadman M, Gowda L, Mirza AS, Abid MB, Hong S, Majhail NS, Kharfan-Dabaja MA, Khurana A, Badar T, Lin Y, Bennani NN, Herr MM, Hu ZH, Wang HL, Baer A, Baro E, Miao H, Spooner C, Xu H, Pasquini MC. Real-world and clinical trial outcomes in large B-cell lymphoma with axicabtagene ciloleucel across race and ethnicity. Blood. 2024 Jun 27;143(26):2722-2734. doi: 10.1182/blood.2023023447. PMID 38635762
- [Derived] Neelapu SS, Jacobson CA, Ghobadi A, Miklos DB, Lekakis LJ, Oluwole OO, Lin Y, Braunschweig I, Hill BT, Timmerman JM, Deol A, Reagan PM, Stiff P, Flinn IW, Farooq U, Goy AH, McSweeney PA, Munoz J, Siddiqi T, Chavez JC, Herrera AF, Bartlett NL, Bot AA, Shen RR, Dong J, Singh K, Miao H, Kim JJ, Zheng Y, Locke FL. Five-year follow-up of ZUMA-1 supports the curative potential of axicabtagene ciloleucel in refractory large B-cell lymphoma. Blood. 2023 May 11;141(19):2307-2315. doi: 10.1182/blood.2022018893. PMID 36821768
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Maloney DG, Kuruvilla J, Liu FF, Kostic A, Kim Y, Bonner A, Zhang Y, Fox CP, Cartron G. Matching-adjusted indirect treatment comparison of liso-cel versus axi-cel in relapsed or refractory large B cell lymphoma. J Hematol Oncol. 2021 Sep 8;14(1):140. doi: 10.1186/s13045-021-01144-9. PMID 34493319
- [Derived] Westin JR, Kersten MJ, Salles G, Abramson JS, Schuster SJ, Locke FL, Andreadis C. Efficacy and safety of CD19-directed CAR-T cell therapies in patients with relapsed/refractory aggressive B-cell lymphomas: Observations from the JULIET, ZUMA-1, and TRANSCEND trials. Am J Hematol. 2021 Oct 1;96(10):1295-1312. doi: 10.1002/ajh.26301. Epub 2021 Aug 13. PMID 34310745
- [Derived] Upadhyay R, Boiarsky JA, Pantsulaia G, Svensson-Arvelund J, Lin MJ, Wroblewska A, Bhalla S, Scholler N, Bot A, Rossi JM, Sadek N, Parekh S, Lagana A, Baccarini A, Merad M, Brown BD, Brody JD. A Critical Role for Fas-Mediated Off-Target Tumor Killing in T-cell Immunotherapy. Cancer Discov. 2021 Mar;11(3):599-613. doi: 10.1158/2159-8290.CD-20-0756. Epub 2020 Dec 17. PMID 33334730
- [Derived] Locke FL, Rossi JM, Neelapu SS, Jacobson CA, Miklos DB, Ghobadi A, Oluwole OO, Reagan PM, Lekakis LJ, Lin Y, Sherman M, Better M, Go WY, Wiezorek JS, Xue A, Bot A. Tumor burden, inflammation, and product attributes determine outcomes of axicabtagene ciloleucel in large B-cell lymphoma. Blood Adv. 2020 Oct 13;4(19):4898-4911. doi: 10.1182/bloodadvances.2020002394. PMID 33035333
- [Derived] Locke FL, Ghobadi A, Jacobson CA, Miklos DB, Lekakis LJ, Oluwole OO, Lin Y, Braunschweig I, Hill BT, Timmerman JM, Deol A, Reagan PM, Stiff P, Flinn IW, Farooq U, Goy A, McSweeney PA, Munoz J, Siddiqi T, Chavez JC, Herrera AF, Bartlett NL, Wiezorek JS, Navale L, Xue A, Jiang Y, Bot A, Rossi JM, Kim JJ, Go WY, Neelapu SS. Long-term safety and activity of axicabtagene ciloleucel in refractory large B-cell lymphoma (ZUMA-1): a single-arm, multicentre, phase 1-2 trial. Lancet Oncol. 2019 Jan;20(1):31-42. doi: 10.1016/S1470-2045(18)30864-7. Epub 2018 Dec 2. PMID 30518502
- [Derived] Neelapu SS, Locke FL, Bartlett NL, Lekakis LJ, Miklos DB, Jacobson CA, Braunschweig I, Oluwole OO, Siddiqi T, Lin Y, Timmerman JM, Stiff PJ, Friedberg JW, Flinn IW, Goy A, Hill BT, Smith MR, Deol A, Farooq U, McSweeney P, Munoz J, Avivi I, Castro JE, Westin JR, Chavez JC, Ghobadi A, Komanduri KV, Levy R, Jacobsen ED, Witzig TE, Reagan P, Bot A, Rossi J, Navale L, Jiang Y, Aycock J, Elias M, Chang D, Wiezorek J, Go WY. Axicabtagene Ciloleucel CAR T-Cell Therapy in Refractory Large B-Cell Lymphoma. N Engl J Med. 2017 Dec 28;377(26):2531-2544. doi: 10.1056/NEJMoa1707447. Epub 2017 Dec 10. PMID 29226797
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KTE-C19-101

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Canada, France, Germany, Israel, Netherlands, and the United States.
Pre-assignment Details: 390 participants were screened. Participants who initially responded and subsequently relapsed, became eligible for second course of conditioning chemotherapy and axicabtagene ciloleucel. Participants received the same axicabtagene ciloleucel regimen as the original target dose.
Groups:
- Phase 1 Study: Axicabtagene Ciloleucel and Conditioning Chemotherapy: Participants with diffuse large B-cell lymphoma (DLBCL), primary mediastinal B-cell lymphoma (PMBCL), or transformed follicular lymphoma (TFL) received conditioning chemotherapy (fludarabine 30 mg/m^2 intravenously [IV] over 30 minutes and cyclophosphamide 500 mg/m^2 IV over 60 minutes) on Days -5, -4, and -3; followed by a single infusion of axicabtagene ciloleucel chimeric antigen receptor (CAR) transduced autologous T cells administered IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of body weight (BW) on Day 0.
- Phase 2 (Pivotal Study): Cohort 1: Participants with refractory DLBCL received conditioning chemotherapy (fludarabine 30 mg/m^2 IV over 30 minutes and cyclophosphamide 500 mg/m^2 IV over 60 minutes) on Days -5, -4, and -3; followed by a single infusion of axicabtagene ciloleucel CAR transduced autologous T cells administered IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of BW on Day 0.
- Phase 2 (Pivotal Study): Cohort 2: Participants with refractory PMBCL or TFL received conditioning chemotherapy (fludarabine 30 mg/m^2 IV over 30 minutes and cyclophosphamide 500 mg/m^2 IV over 60 minutes) on Days -5, -4, and -3; followed by a single infusion of axicabtagene ciloleucel CAR transduced autologous T cells administered IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of BW on Day 0.
- Phase 2 (Safety Management Study): Cohort 3: Participants with relapsed or refractory transplant ineligible DLBCL, PMBCL, or TFL received conditioning chemotherapy (fludarabine 30 mg/m^2 IV over 30 minutes and cyclophosphamide 500 mg/m^2 IV over 60 minutes) on Days -5, -4, and -3; followed by a single infusion of axicabtagene ciloleucel CAR transduced autologous T cells administered IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of BW on Day 0. Participants also received a prophylactic regimen of levetiracetam (750 mg orally or IV twice daily (BID) starting on Day 0) and tocilizumab (8 mg/kg IV over 1 hour (not to exceed 800 mg)) on Day 2).
- Phase 2 (Safety Management Study): Cohort 4: Participants with r/r DLBCL, PMBCL ,TFL, or high-grade B-cell lymphoma (HGBCL) after 2 systemic lines of therapy received optional bridging therapy (dexamethasone 20mg to 40mg,either orally or IV daily for 1 to 4 days or 1g/m^2 of high-dose methylprednisolone(HDMP) for 3 days with rituximab at 375mg/m^2 weekly for 3 weeks or bendamustine 90 mg/m^2 on Days 1 and 2 and rituximab 375mg/m^2 on Day 1), conditioning chemotherapy (fludarabine 30mg/m^2 IV and cyclophosphamide 500mg/m^2 IV)on Days -5,-4, and -3; followed by single infusion of axicabtagene ciloleucel CAR transduced autologous T cells IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of BW. Participants also received a prophylactic regimen of levetiracetam (750 mg orally or IV twice daily (BID) starting on Day 0). Participants received tocilizumab (initiated on persistent Grade 1 cytokine release syndrome (CRS) for over 24 hours) and dexamethasone (persistent Grade 1 CRS for over 72 hours and at onset of Grade 1 neurologic toxicity).
- Phase 2 (Safety Management Study): Cohort 5: Participants with r/r DLBCL, PMBCL ,TFL, or HGBCL after 2 systemic lines of therapy received debulking therapy (R-CHOP:rituximab 375mg/m^2 D1,doxorubicin 50mg/m^2 D1,prednisone 100mg D1 to D5,cyclophosphamide 750mg/m^2 D1,vincristine 1.4 mg/m^2 D1 or R-ICE:rituximab 375mg/ m^2 D1,ifosfamide 5g/m^2 24h-CI D2,carboplatin AUC5 D2 maximum dose 800mg,etoposide 100 mg/m^2/day D1 to D3 or R-GEMOX:rituximab 375mg/m^2 D1,gemcitabine 1000mg/m^2 D2,oxaliplatin 100mg/m^2 D2 or R-GDP:rituximab 375mg/m^2 D1 or D8,gemcitabine 1g/m^2 D1 & D8,dexamethasone 40mg D1 to D4,cisplatin 75mg/m^2 D1(or carboplatin AUC5 D1) or radiotherapy:20 to 30 Gy), conditioning chemotherapy (fludarabine 30mg/m^2 IV and cyclophosphamide 500mg/m^2 IV)on Days -5,-4, and -3; followed by single infusion of axicabtagene ciloleucel at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of BW on Day 0. Participants also received a prophylactic regimen of levetiracetam (750 mg orally or IV BID starting on D0).D=Day.
- Phase 2 (Safety Management Study): Cohort 6: Participants with r/r DLBCL, PMBCL ,TFL, or HGBCL after 2 systemic lines of therapy may have received bridging therapy (dexamethasone 20mg to 40mg, either orally or IV daily for 1 to 4 days or 1g/m^2 of high-dose methylprednisolone(HDMP) for 3 days with rituximab at 375mg/m^2 weekly for 3 weeks or bendamustine 90 mg/m^2 on Days 1 and 2 and rituximab 375mg/m^2 on Day 1), conditioning chemotherapy (fludarabine 30mg/m^2 IV and cyclophosphamide 500mg/m^2 IV)on Days -5,-4, and -3; followed by single infusion of axicabtagene ciloleucel CAR transduced autologous T cells IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of BW on Day 0. Participants also received a prophylactic regimen of levetiracetam (750 mg orally or IV twice daily (BID) starting on Day 0) and corticosteroids (dexamethasone, 10 mg once daily on Days 0, 1, and 2). Participants received tocilizumab (initiated on persistent Grade 1 CRS for over 24 hours) and dexamethasone (persistent Grade 1 CRS for over 72 hours and at onset of Grade 1 neurologic toxicity).
Period: Overall Study
Arm/Group | Phase 1 Study: Axicabtagene Ciloleucel and Conditioning Chemotherapy | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2 | Phase 2 (Safety Management Study): Cohort 3 | Phase 2 (Safety Management Study): Cohort 4 | Phase 2 (Safety Management Study): Cohort 5 | Phase 2 (Safety Management Study): Cohort 6
Started | 8 | 81 | 30 | 42 | 46 | 58 | 42
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 81 | 30 | 42 | 46 | 58 | 42
Not completed — Death | 5 | 53 | 11 | 20 | 16 | 32 | 17
Not completed — Full consent withdrawal | 0 | 0 | 0 | 1 | 3 | 0 | 3
Not completed — Lost to Follow-up | 0 | 5 | 2 | 0 | 1 | 1 | 1
Not completed — Enrolled but did not initiate axicabtagene ciloleucel | 1 | 4 | 6 | 4 | 5 | 8 | 2
Not completed — Reason not specified | 2 | 19 | 11 | 17 | 21 | 17 | 19

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants treated with any dose of axicabtagene ciloleucel.
Groups:
- Phase 2 (Safety Management Study): Cohort 4: Participants with r/r DLBCL, PMBCL ,TFL, or high-grade B-cell lymphoma (HGBCL) after 2 systemic lines of therapy received optional bridging therapy (dexamethasone 20mg to 40mg,either orally or IV daily for 1 to 4 days or 1g/m^2 of high-dose methylprednisolone(HDMP) for 3 days with rituximab at 375mg/m^2 weekly for 3 weeks or bendamustine 90 mg/m^2 on Days 1 and 2 and rituximab 375mg/m^2 on Day 1), conditioning chemotherapy (fludarabine 30mg/m^2 IV and cyclophosphamide 500mg/m^2 IV)on Days -5,-4, and -3; followed by single infusion of axicabtagene ciloleucel CAR transduced autologous T cells IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg of BW. Participants also received a prophylactic regimen of levetiracetam (750 mg orally or IV twice daily (BID) starting on Day 0). Participants received tocilizumab (initiated on persistent Grade 1 CRS for over 24 hours) and dexamethasone (persistent Grade 1 CRS for over 72 hours and at onset of Grade 1 neurologic toxicity).
- Total: Total of all reporting groups
Arm/Group | Phase 1 Study: Axicabtagene Ciloleucel and Conditioning Chemotherapy | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2 | Phase 2 (Safety Management Study): Cohort 3 | Phase 2 (Safety Management Study): Cohort 4 | Phase 2 (Safety Management Study): Cohort 5 | Phase 2 (Safety Management Study): Cohort 6 | Total
Number analyzed (Participants) | 7 | 77 | 24 | 38 | 41 | 50 | 40 | 277
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 60 | 17 | 30 | 28 | 35 | 20 | 194
  >=65 years | 3 | 17 | 7 | 8 | 13 | 15 | 20 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (17.5) | 57 (10.6) | 53 (15.5) | 51 (13.0) | 57 (12.9) | 58 (9.9) | 64 (9.4) | 57 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 27 | 6 | 17 | 13 | 14 | 17 | 96
  Male | 5 | 50 | 18 | 21 | 28 | 36 | 23 | 181
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 16 | 2 | 5 | 0 | 1 | 2 | 27
  Not Hispanic or Latino | 6 | 61 | 22 | 33 | 40 | 49 | 38 | 249
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 5 | 69 | 18 | 31 | 33 | 33 | 34 | 223
  Race: Other or More Than One Race | 1 | 5 | 2 | 3 | 8 | 10 | 5 | 34
  Race: Black or African American | 1 | 3 | 1 | 3 | 0 | 2 | 1 | 11
  Race: Asian | 0 | 0 | 3 | 1 | 0 | 5 | 0 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 0 | 0 | 1 | 7 | 15 | 0 | 23
  France | 0 | 0 | 0 | 0 | 9 | 13 | 8 | 30
  Germany | 0 | 0 | 0 | 0 | 12 | 9 | 0 | 21
  Israel | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 6
  Netherlands | 0 | 0 | 0 | 5 | 11 | 13 | 6 | 35
  United States | 7 | 77 | 23 | 30 | 0 | 0 | 25 | 162

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 Study: Number of Participants Experiencing Adverse Events (AEs) Defined as Dose Limiting Toxicities (DLTs)
Description: DLT was defined as axicabtagene ciloleucel-related events with onset within first 30 days following infusion:
  * Grade (GR) 4 neutropenia lasting > 21 days and GR 4 thrombocytopenia lasting > 35 days from day of cell transfer;
  * Any axicabtagene ciloleucel-related AE requiring intubation;
  * All other GR 3 toxicities lasting > 3 days and all GR 4 toxicities, with exception of following conditions which were not considered DLTs: aphasia/dysphasia or confusion/cognitive disturbance which resolved to GR ≤ 1 within 2 weeks and to baseline within 4 weeks; fever GR 3; myelosuppression defined as lymphopenia, decreased hemoglobin, neutropenia and thrombocytopenia unless neutropenia and thrombocytopenia met DLT definition described above; immediate hypersensitivity reactions occurring within 2 hours of cell infusion that were reversible to a ≤ GR 2 within 24 hours of cell administration with standard therapy; hypogammaglobulinemia GR 3 or 4.
Time Frame: First infusion date of axicabtagene ciloleucel up to 30 days
Population: DLT-Evaluable Analysis Set included participants treated in Phase 1 dosing cohort who received the target dose and were followed for at least 30 days after the axicabtagene ciloleucel infusion; or dose of anti-CD19 CAR T cells (axicabtagene ciloleucel) lower than the target for that cohort and experienced a DLT during the 30 day post-infusion period.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Study: Axicabtagene Ciloleucel and Conditioning Chemotherapy
Number analyzed (Participants) | 6
Participants | 1

2. Primary Outcome: Phase 2 Pivotal Study (Cohorts 1 and 2): Overall Response Rate (ORR) as Assessed by Investigator Per Revised International Working Group (IWG) Response Criteria for Malignant Lymphoma
Description: ORR was defined as the percentage of participants achieving either a complete response (CR) or a partial response (PR), as assessed by the study investigators using revised IWG Response Criteria for Malignant Lymphoma (Cheson et al, 2007). CR: complete disappearance of all detectable clinical evidence of disease and disease-related symptoms; all lymph nodes and nodal masses must have regressed to normal size; spleen and/or liver must be normal size, not be palpable, and no nodules; bone marrow aspirate and biopsy must show no evidence of disease. PR: a ≥ 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses; no increase in size of nodes, liver or spleen and no new sites of disease; multiple splenic and hepatic nodules (if present) must regress by ≥ 50% in the SPD; > 50% decrease in the greatest transverse diameter for single nodules. 95% confidence interval (CI) was calculated by Clopper-Pearson method.
Time Frame: First infusion date of axicabtagene ciloleucel up to last follow-up visit (maximum duration: 7.7 years)
Population: The Modified Intent-to-Treat (mITT) analysis set included all participants treated with at least 1.0 x 10^6 anti-CD19 CAR T cells/kg.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2
Number analyzed (Participants) | 77 | 24
percentage of participants | 83 [73 to 91] | 83 [63 to 95]

3. Primary Outcome: Phase 2 Safety Management Study (Cohort 3): Percentage of Participants With Treatment-Emergent Cytokine Release Syndrome (CRS) and Neurologic Toxicities by Severity Grades
Description: TEAE was defined as any AE with onset on or after the start of treatment. CRS events were graded by Lee et al 2014. Grade 1 : No life threatening symptoms and require symptomatic treatment only; Grade 2: Symptoms require and respond to moderate intervention; Grade 3: Symptoms require and respond to aggressive intervention; Grade 4: Life-threatening symptoms and requirements for ventilator support or continuous venovenous hemodialysis (CVVHD), and Grade 5: Death. Neurologic toxicities were graded by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Grade 1: Mild, asymptomatic or mild symptoms and intervention not indicated; Grade 2: Moderate and minimal, local or noninvasive intervention indicated; Grade 3: Severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated; Grade 4: Life-threatening and urgent intervention indicated; Grade 5: Death related to AE.
Time Frame: First infusion date of axicabtagene ciloleucel up to last follow-up visit (maximum duration: 6.8 years)
Population: The Safety Analysis Set included all participants treated with any dose of axicabtagene ciloleucel.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 (Safety Management Study): Cohort 3
Number analyzed (Participants) | 38
percentage of participants
  Worst Grade 1 CRS | 34
  Worst Grade 2 CRS | 55
  Worst Grade 3 CRS | 0
  Worst Grade 4 CRS | 3
  Worst Grade 5 CRS | 0
  Worst Grade ≥ 3 CRS | 3
  Worst Grade 1 Neurologic Toxicities | 24
  Worst Grade 2 Neurologic Toxicities | 21
  Worst Grade 3 Neurologic Toxicities | 37
  Worst Grade 4 Neurologic Toxicities | 3
  Worst Grade 5 Neurologic Toxicities | 3
  Worst Grade ≥ 3 Neurologic Toxicities | 42

4. Primary Outcome: Phase 2 Safety Management Study (Cohort 4): Percentage of Participants With Treatment-Emergent CRS and Neurologic Toxicities by Severity Grades
Description: TEAE was defined as any AE with onset on or after the start of treatment. CRS events were graded by Lee et al 2014. Grade 1 : No life threatening symptoms and require symptomatic treatment only; Grade 2: Symptoms require and respond to moderate intervention; Grade 3: Symptoms require and respond to aggressive intervention; Grade 4: Life-threatening symptoms and requirements for ventilator support or CVVHD, and Grade 5: Death. Neurologic toxicities were graded by CTCAE version 4.03. Grade 1: Mild, asymptomatic or mild symptoms and intervention not indicated; Grade 2: Moderate and minimal, local or noninvasive intervention indicated; Grade 3: Severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated; Grade 4: Life-threatening and urgent intervention indicated; Grade 5: Death related to AE.
Time Frame: First infusion date of axicabtagene ciloleucel up to last follow-up visit (maximum duration: 5.4 years)
Population: The Safety Analysis Set included all participants treated with any dose of axicabtagene ciloleucel.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 (Safety Management Study): Cohort 4
Number analyzed (Participants) | 41
percentage of participants
  Worst Grade 1 CRS | 32
  Worst Grade 2 CRS | 59
  Worst Grade 3 CRS | 2
  Worst Grade 4 CRS | 0
  Worst Grade 5 CRS | 0
  Worst Grade ≥ 3 CRS | 2
  Worst Grade 1 Neurologic Toxicities | 34
  Worst Grade 2 Neurologic Toxicities | 10
  Worst Grade 3 Neurologic Toxicities | 17
  Worst Grade 4 Neurologic Toxicities | 0
  Worst Grade 5 Neurologic Toxicities | 0
  Worst Grade ≥ 3 Neurologic Toxicities | 17

5. Primary Outcome: Phase 2 Safety Management Study (Cohort 5): Percentage of Participants With Treatment-Emergent CRS and Neurologic Toxicities by Severity Grades
Description: as for outcome 4
Time Frame: First infusion date of axicabtagene ciloleucel up to last follow-up visit (maximum duration: 4.4 years)
Population: The Safety Analysis Set included all participants treated with any dose of axicabtagene ciloleucel.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 (Safety Management Study): Cohort 5
Number analyzed (Participants) | 50
percentage of participants
  Worst Grade 1 CRS | 38
  Worst Grade 2 CRS | 46
  Worst Grade 3 CRS | 0
  Worst Grade 4 CRS | 2
  Worst Grade 5 CRS | 0
  Worst Grade ≥ 3 CRS | 2
  Worst Grade 1 Neurologic Toxicities | 26
  Worst Grade 2 Neurologic Toxicities | 18
  Worst Grade 3 Neurologic Toxicities | 10
  Worst Grade 4 Neurologic Toxicities | 2
  Worst Grade 5 Neurologic Toxicities | 0
  Worst Grade ≥ 3 Neurologic Toxicities | 12

6. Primary Outcome: Phase 2 Safety Management Study (Cohort 6): Percentage of Participants With Treatment-Emergent CRS and Neurologic Toxicities by Severity Grades
Description: as for outcome 4
Time Frame: First infusion date of axicabtagene ciloleucel up to last follow-up visit (maximum duration: 4.1 years)
Population: The Safety Analysis Set included all participants treated with any dose of axicabtagene ciloleucel.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 (Safety Management Study): Cohort 6
Number analyzed (Participants) | 40
percentage of participants
  Worst Grade 1 CRS | 35
  Worst Grade 2 CRS | 45
  Worst Grade 3 CRS | 0
  Worst Grade 4 CRS | 0
  Worst Grade 5 CRS | 0
  Worst Grade ≥ 3 CRS | 0
  Worst Grade 1 Neurologic Toxicities | 23
  Worst Grade 2 Neurologic Toxicities | 18
  Worst Grade 3 Neurologic Toxicities | 8
  Worst Grade 4 Neurologic Toxicities | 5
  Worst Grade 5 Neurologic Toxicities | 5
  Worst Grade ≥ 3 Neurologic Toxicities | 18

7. Secondary Outcome: Phase 2: Duration of Response (DOR) as Assessed by Investigator Per Revised IWG Response Criteria for Malignant Lymphoma
Description: Among participants who experience an objective response (OR), DOR was defined as the date of their first objective response (CR or PR which was subsequently confirmed) to disease progression per the revised IWG Response Criteria for Malignant Lymphoma or death regardless of cause. CR and PR as defined in outcome measure 2. Disease progression (PD) was defined by at least one of the following: ≥ 50% increase from nadir in the sum of the products of at least 2 lymph nodes, or at least a 50% increase in the product of the diameters of a single lymph node; appearance of a new lesion > 1.5 cm in any axis; ≥ 50% increase in size of splenic or hepatic nodules; ≥ 50% increase in the longest diameter of any single previously identified node > 1 cm in its short axis. Kaplan-Meier (KM) estimates was used for analyses.
Time Frame: First OR to last follow-up visit (maximum duration: 7.7, 6.8, 5.4, 4.4, 4.1 years for Cohorts 1, 2, 3, 4, 5, and 6 respectively)
Population: Participants in the mITT Analysis Set with objective response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2 | Phase 2 (Safety Management Study): Cohort 3 | Phase 2 (Safety Management Study): Cohort 4 | Phase 2 (Safety Management Study): Cohort 5 | Phase 2 (Safety Management Study): Cohort 6
Number analyzed (Participants) | 64 | 20 | 24 | 31 | 36 | 38
months | 5.0 [2.1 to 34.7] | 75.4 [11.1 to NA] — Upper limit of 95% CI was not estimable because almost 50% of participants were censored. | NA [5.0 to NA] — Median and upper limit of 95% CI was not estimable because almost 50% of participants were censored. | NA [NA to NA] — Median and upper and lower limit of 95% CI was not estimable because almost 50% of participants were censored. | 27.5 [2.2 to NA] — Upper limit of 95% CI was not estimable because almost 50% of participants were censored. | NA [7.8 to NA] — Median and upper limit of 95% CI was not estimable because almost 50% of participants were censored.

8. Secondary Outcome: Phase 1 Study: ORR as Assessed by Investigator Per Revised IWG Response Criteria for Malignant Lymphoma
Description: ORR was defined as the percentage of participants achieving either a CR or a PR, as assessed by the study investigators using revised IWG Response Criteria for Malignant Lymphoma (Cheson et al, 2007). CR: complete disappearance of all detectable clinical evidence of disease and disease-related symptoms; all lymph nodes and nodal masses must have regressed to normal size; spleen and/or liver must be normal size, not be palpable, and no nodules; bone marrow aspirate and biopsy must show no evidence of disease. PR: a ≥ 50% decrease in SPD of up to 6 of the largest dominant nodes or nodal masses; no increase in size of nodes, liver or spleen and no new sites of disease; multiple splenic and hepatic nodules (if present) must regress by ≥ 50% in the SPD; > 50% decrease in the greatest transverse diameter for single nodules.
Time Frame: First infusion date of axicabtagene ciloleucel to the data cutoff date of 27 January 2017 (maximum: 20 months)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 Study: Axicabtagene Ciloleucel and Conditioning Chemotherapy
Number analyzed (Participants) | 7
percentage of participants | 71

9. Secondary Outcome: Phase 2 Pivotal Study (Cohorts 1 and 2): ORR Per Independent Radiological Review Committee (IRRC)
Description: ORR was defined as the percentage of participants achieving either a CR or a PR, as assessed by the IRRC using revised IWG Response Criteria for Malignant Lymphoma. CR: complete disappearance of all detectable clinical evidence of disease and disease-related symptoms; all lymph nodes and nodal masses must have regressed to normal size; spleen and/or liver must be normal size, not be palpable, and no nodules; bone marrow aspirate and biopsy must show no evidence of disease. PR: a ≥ 50% decrease in SPD of up to 6 of the largest dominant nodes or nodal masses; no increase in size of nodes, liver or spleen and no new sites of disease; multiple splenic and hepatic nodules (if present) must regress by ≥ 50% in the SPD; > 50% decrease in the greatest transverse diameter for single nodules. 95% CI was calculated by Clopper-Pearson method.
Time Frame: First infusion date of axicabtagene ciloleucel to the data cutoff date of 11 August 2018 (maximum: 2.7 years)
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2
Number analyzed (Participants) | 77 | 24
percentage of participants | 70 [59 to 80] | 88 [68 to 97]

10. Secondary Outcome: Phase 2 Safety Management Study (Cohorts 3, 4, 5, and 6): ORR as Assessed by Investigator Per the Revised IWG Response Criteria for Malignant Lymphoma
Description: ORR was defined as the percentage of participants achieving either a CR or a PR, as assessed by the study investigators using revised IWG Response Criteria for Malignant Lymphoma (Cheson et al, 2007). CR: complete disappearance of all detectable clinical evidence of disease and disease-related symptoms; all lymph nodes and nodal masses must have regressed to normal size; spleen and/or liver must be normal size, not be palpable, and no nodules; bone marrow aspirate and biopsy must show no evidence of disease. PR: a ≥ 50% decrease in SPD of up to 6 of the largest dominant nodes or nodal masses; no increase in size of nodes, liver or spleen and no new sites of disease; multiple splenic and hepatic nodules (if present) must regress by ≥ 50% in the SPD; > 50% decrease in the greatest transverse diameter for single nodules. 95% CI was calculated by Clopper-Pearson method.
Time Frame: First infusion date of axicabtagene ciloleucel to last follow-up visit (maximum duration: 6.8, 5.4, 4.4, 4.1 years for Cohorts 3, 4, 5, and 6 respectively)
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 (Safety Management Study): Cohort 3 | Phase 2 (Safety Management Study): Cohort 4 | Phase 2 (Safety Management Study): Cohort 5 | Phase 2 (Safety Management Study): Cohort 6
Number analyzed (Participants) | 38 | 41 | 50 | 40
percentage of participants | 63 [46 to 78] | 76 [60 to 88] | 72 [58 to 84] | 95 [83 to 99]

11. Secondary Outcome: Phase 2: Progression-Free Survival (PFS) as Assessed by Investigator Per Revised IWG Response Criteria for Malignant Lymphoma
Description: PFS was defined as the time from the axicabtagene ciloleucel infusion date to the date of disease progression per the revised IWG Response Criteria for Malignant Lymphoma (Cheson et al, 2007) or death from any cause. Participants not meeting the criteria for progression by the analysis data cutoff date were censored at their last evaluable disease assessment date. Disease progression was defined by at least one of the following: ≥ 50% increase from nadir in the sum of the products of at least 2 lymph nodes, or at least a 50% increase in the product of the diameters of a single lymph node; appearance of a new lesion > 1.5 cm in any axis; ≥ 50% increase in size of splenic or hepatic nodules; ≥ 50% increase in the longest diameter of any single previously identified node > 1 cm in its short axis. KM estimates was used for analyses.
Time Frame: First infusion date of axicabtagene ciloleucel to disease progression or death regardless of cause (maximum duration: 7.7, 6.8, 5.4, 4.4, 4.1 years for Cohorts 1, 2, 3, 4, 5, and 6 respectively)
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2 | Phase 2 (Safety Management Study): Cohort 3 | Phase 2 (Safety Management Study): Cohort 4 | Phase 2 (Safety Management Study): Cohort 5 | Phase 2 (Safety Management Study): Cohort 6
Number analyzed (Participants) | 77 | 24 | 38 | 41 | 50 | 40
months | 5.1 [3.0 to 8.8] | 49.1 [3.7 to NA] — Upper limit of 95% CI was not estimable because almost 50% of participants were censored. | 6.2 [2.4 to NA] — Upper limit of 95% CI was not estimable because almost 50% of participants were censored. | NA [3.0 to NA] — Median and upper limit of 95% CI was not estimable because almost 50% of participants were censored. | 3.1 [2.9 to 29.1] | NA [8.7 to NA] — Median and upper limit of 95% CI was not estimable because almost 50% of participants were censored.

12. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as the time from axicabtagene ciloleucel infusion to the date of death. Participants who did not die by the analysis data cutoff date were censored at their last contact date. KM estimates was used for analyses.
Time Frame: First infusion date of axicabtagene ciloleucel to the date of death regardless of cause (maximum duration: 7.7, 6.8, 5.4, 4.4, 4.1 years for Cohorts 1, 2, 3, 4, 5, and 6 respectively)
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2 | Phase 2 (Safety Management Study): Cohort 3 | Phase 2 (Safety Management Study): Cohort 4 | Phase 2 (Safety Management Study): Cohort 5 | Phase 2 (Safety Management Study): Cohort 6
Number analyzed (Participants) | 77 | 24 | 38 | 41 | 50 | 40
months | 15.4 [10.4 to 45.7] | NA [15.0 to NA] — Median and upper limit of 95% CI was not estimable because almost 50% of participants were censored. | 34.8 [5.4 to NA] — Upper limit of 95% CI was not estimable because almost 50% of participants were censored. | NA [14.6 to NA] — Median and upper limit of 95% CI was not estimable because almost 50% of participants were censored. | 20.6 [12.6 to 43.1] | NA [18.9 to NA] — Median and upper limit of 95% CI was not estimable because almost 50% of participants were censored.

13. Secondary Outcome: Phase 2 Pivotal Study (Cohorts 1 and 2): Duration of Response (DOR) Using IRRC Per Cheson 2007
Description: Among participants who experience an objective response, DOR was defined as the date of their first objective response (CR or PR which was subsequently confirmed) to PD, as assessed by the IRRC using revised IWG Response Criteria for Malignant Lymphoma (Cheson et al, 2007) or death regardless of cause. CR and PR as defined in outcome measure 2. PD was defined by at least one of the following: ≥ 50% increase from nadir in the sum of the products of at least 2 lymph nodes, or at least a 50% increase in the product of the diameters of a single lymph node; appearance of a new lesion > 1.5 cm in any axis; ≥ 50% increase in size of splenic or hepatic nodules; ≥ 50% increase in the longest diameter of any single previously identified node > 1 cm in its short axis. Kaplan-Meier (KM) estimates was used for analyses.
Time Frame: First objective response up to the data cutoff date of 11 August 2018 (maximum: 2.7 years)
Population: Participants in the mITT Analysis Set with objective response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2
Number analyzed (Participants) | 54 | 21
months | NA [5.4 to NA] — Median and upper limit of 95% CI was not estimable because almost 50% of participants were censored. | NA [11.1 to NA] — Median and upper limit of 95% CI was not estimable because almost 50% of participants were censored.

14. Secondary Outcome: Phase 2 Pivotal Study (Cohorts 1 and 2): Best Overall Response Using IRRC Per Cheson 2007
Description: The best overall response for each participant was based on the assessments of response (CR, PR, stable disease [SD], PD, and not done [ND]) made by the the IRRC using IWG 2007 criteria (Cheson et al, 2007). CR and PR as defined in outcome measure 2. PD defined by at least one of the following: ≥ 50% increase from nadir in the sum of the products of at least 2 lymph nodes, or at least a 50% increase in the product of the diameters of a single lymph node; appearance of a new lesion > 1.5 cm in any axis; ≥ 50% increase in size of splenic or hepatic nodules; ≥ 50% increase in the longest diameter of any single previously identified node > 1 cm in its short axis. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Percentage of participants with best overall response of CR, PR, SD, PD, and ND was reported.
Time Frame: First infusion date of axicabtagene ciloleucel to the data cutoff date of 11 August 2018 (maximum: 2.7 years)
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2
Number analyzed (Participants) | 77 | 24
percentage of participants
  CR | 51 | 67
  PR | 19 | 21
  SD | 21 | 4
  PD | 8 | 4
  ND | 1 | 4

15. Secondary Outcome: Phase 2 Pivotal Study (Cohorts 1 and 2): PFS Using IRRC Per Cheson 2007
Description: PFS was defined as the time from the axicabtagene ciloleucel infusion date to the date of disease progression as assessed by the IRRC using revised IWG Response Criteria for Malignant Lymphoma (Cheson et al, 2007) or death from any cause. Participants not meeting the criteria for progression by the analysis data cutoff date were censored at their last evaluable disease assessment date. PD defined by at least one of the following: ≥ 50% increase from nadir in the sum of the products of at least 2 lymph nodes, or at least a 50% increase in the product of the diameters of a single lymph node; appearance of a new lesion > 1.5 cm in any axis; ≥ 50% increase in size of splenic or hepatic nodules; ≥ 50% increase in the longest diameter of any single previously identified node > 1 cm in its short axis. KM estimates was used for analyses.
Time Frame: First infusion date of axicabtagene ciloleucel to the data cutoff date of 11 August 2018 (maximum: 2.7 years)
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2
Number analyzed (Participants) | 77 | 24
months | 6.9 [4.5 to 15.0] | NA [9.0 to NA] — Median and upper limit of 95% CI was not estimable because almost 50% of participants were censored.

16. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event was defined as any untoward medical occurrence in a clinical trial participants. The event did not necessarily have a relationship with study treatment. Adverse events included worsening of a pre-existing medical condition. Worsening indicated that the pre-existing medical condition had increased in severity, frequency, and/or duration or had an association with a worse outcome. A pre-existing condition that had not worsened during the study or involved an intervention such as elective cosmetic surgery or a medical procedure while on study, was not considered an adverse event. TEAE was defined as any AE with onset on or after the start of treatment.
Time Frame: First infusion date of axicabtagene ciloleucel up to last follow up visit (maximum duration: 7.7 years)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 Study: Axicabtagene Ciloleucel and Conditioning Chemotherapy | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2 | Phase 2 (Safety Management Study): Cohort 3 | Phase 2 (Safety Management Study): Cohort 4 | Phase 2 (Safety Management Study): Cohort 5 | Phase 2 (Safety Management Study): Cohort 6
Number analyzed (Participants) | 7 | 77 | 24 | 38 | 41 | 50 | 40
percentage of participants | 100 | 100 | 100 | 100 | 100 | 100 | 100

17. Secondary Outcome: Percentage of Participants With Clinically Significant Changes in Laboratory Values Reported as Grade 3 or Higher TEAEs
Description: Grading categories were determined by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Grade 1: mild, Grade 2: moderate, Grade 3: severe or medically significant, Grade 4: life-threatening.
Time Frame: First infusion date of axicabtagene ciloleucel up to last follow up visit (maximum duration: 7.7 years)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 Study: Axicabtagene Ciloleucel and Conditioning Chemotherapy | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2 | Phase 2 (Safety Management Study): Cohort 3 | Phase 2 (Safety Management Study): Cohort 4 | Phase 2 (Safety Management Study): Cohort 5 | Phase 2 (Safety Management Study): Cohort 6
Number analyzed (Participants) | 7 | 77 | 24 | 38 | 41 | 50 | 40
percentage of participants | 100 | 96 | 96 | 97 | 98 | 100 | 100

18. Secondary Outcome: Percentage of Participants With Anti-Axicabtagene Ciloleucel Antibodies
Time Frame: First infusion date of axicabtagene ciloleucel up to last follow-up visit (maximum duration: 7.7, 6.8, 5.4, 4.4, 4.1 years for Phase 1 and Phase 2 Cohorts 1, 2, 3, 4, 5, and 6 respectively)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 Study: Axicabtagene Ciloleucel and Conditioning Chemotherapy | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2 | Phase 2 (Safety Management Study): Cohort 3 | Phase 2 (Safety Management Study): Cohort 4 | Phase 2 (Safety Management Study): Cohort 5 | Phase 2 (Safety Management Study): Cohort 6
Number analyzed (Participants) | 7 | 77 | 24 | 38 | 41 | 50 | 40
percentage of participants | 29 | 5 | 8 | 11 | 0 | 8 | 8

19. Secondary Outcome: Pharmacokinetics: Peak Level of Anti-CD19 CAR T Cells in Blood
Description: Peak was defined as the maximum number of CAR T cells measured post-infusion.
Time Frame: Baseline up to Month 60 (for Phase 1 and Phase 2 Cohorts 1, 2, and 3); Baseline up to Month 24 (for Phase 2 Cohorts 4, 5, and 6)
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: cells/µL
Arm/Group | Phase 1 Study: Axicabtagene Ciloleucel and Conditioning Chemotherapy | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2 | Phase 2 (Safety Management Study): Cohort 3 | Phase 2 (Safety Management Study): Cohort 4 | Phase 2 (Safety Management Study): Cohort 5 | Phase 2 (Safety Management Study): Cohort 6
Number analyzed (Participants) | 6 | 76 | 22 | 36 | 39 | 49 | 40
cells/µL | 58.512 [18.028 to 147.732] | 31.512 [12.445 to 74.746] | 58.633 [27.884 to 103.190] | 53.670 [22.813 to 146.075] | 52.91 [27.25 to 92.78] | 26.63 [12.52 to 117.53] | 64.38 [6.27 to 131.24]

20. Secondary Outcome: Pharmacodynamics: Peak Level of Cytokines in Serum (Phase 1 and Phase 2 Cohorts 1, 2, and 3)
Description: Peak was defined as the maximum post-baseline level of the cytokine. Following key cytokines were measured: interferon-gamma induced protein 10 (IP-10), ferritin, granzyme B, intercellular adhesion molecule (ICAM-1), interferon-gamma (IFN-gamma), interleukin-1 receptor antagonist (IL-1RA), IL-2, interleukin-2 receptor alpha (IL-2 R alpha), IL-6, IL-7, IL-8, IL-10, IL-15, perforin, tumor necrosis factor alpha (TNF alpha), and vascular cell adhesion molecule- 1 (VCAM-1).
Time Frame: Baseline up to Month 3
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 1 Study: Axicabtagene Ciloleucel and Conditioning Chemotherapy | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2 | Phase 2 (Safety Management Study): Cohort 3
Number analyzed (Participants) | 7 | 77 | 24 | 38
pg/mL
  IP-10 | 2000.0 [147.0 to 2000.0] | 2000.0 [628.1 to 2000.0] | 2000.0 [434.2 to 2000.0] | 2000.0 [541.0 to 2000.0]
  Granzyme B | 33.1 [0.6 to 463.8] | 31.1 [1.0 to 3306.0] | 17.3 [1.0 to 406.8] | 44.1 [1.0 to 534.6]
  ICAM-1 | 792754.3 [537796.8 to 2424877.7] | 1322829.3 [557025.0 to 7495123.2] | 989188.4 [544589.3 to 4588974.8] | 1009966.4 [256768.6 to 4879749.7]
  IFN-gamma | 792.0 [81.1 to 1876.0] | 493.8 [32.4 to 1876.0] | 364.9 [7.5 to 1876.0] | 1857.2 [65.0 to 1876.0]
  IL-1 RA | 2173.3 [544.3 to 4000.0] | 2371.2 [510.8 to 4000.0] | 1999.9 [649.9 to 4000.0] | 2160.5 [653.7 to 4000.0]
  IL-2 | 18.4 [3.1 to 91.0] | 25.0 [0.9 to 123.1] | 13.4 [0.9 to 63.7] | 20.0 [0.9 to 189.4]
  IL-2 R alpha | 16872.7 [2189.0 to 34044.5] | 14383.7 [78.0 to 100000.0] | 7817.3 [78.0 to 66024.6] | 12386.4 [3002.6 to 100000.0]
  IL-6 | 305.3 [2.4 to 976.0] | 89.4 [3.5 to 976.0] | 44.6 [3.6 to 976.0] | 921.8 [13.3 to 976.0]
  IL-7 | 51.5 [31.2 to 71.5] | 38.9 [13.8 to 153.5] | 44.1 [27.9 to 98.8] | 38.8 [19.1 to 83.8]
  IL-8 | 86.4 [17.1 to 750.0] | 118.4 [14.2 to 750.0] | 77.2 [9.8 to 750.0] | 120.9 [10.3 to 750.0]
  IL-10 | 52.5 [3.8 to 614.0] | 43.9 [0.7 to 466.0] | 18.8 [0.7 to 263.6] | 48.2 [1.8 to 466.0]
  IL-15 | 57.1 [18.7 to 271.3] | 56.5 [13.1 to 226.6] | 47.6 [11.3 to 195.2] | 50.3 [21.9 to 537.3]
  Perforin | 5389.0 [2582.7 to 20724.3] | 11309.5 [2282.3 to 39818.9] | 8278.7 [2332.6 to 31857.7] | 15411.9 [4327.4 to 30575.9]
  TNF alpha | 10.5 [1.8 to 443.1] | 8.6 [2.6 to 166.9] | 6.8 [2.2 to 44.9] | 10.9 [3.3 to 52.1]
  VCAM-1 | 1387033.6 [609223.2 to 8424222.9] | 1478356.8 [642372.6 to 3859375.8] | 1058453.9 [634769.7 to 2864040.2] | 1367940.7 [721050.0 to 5184238.4]

21. Secondary Outcome: Pharmacodynamics: Peak Level of Cytokines (IP-10, Granzyme B, IFN-gamma, IL-1 RA, IL-10, IL-15, IL-2, IL-6, IL-7, IL-8, TNF Alpha, and GM-CSF) in Serum (Phase 2 Cohorts 4, 5, and 6)
Description: Peak was defined as the maximum post-baseline level of the cytokine. Following key cytokines were measured: IP-10, granzyme B, IFN-gamma, IL-1 RA, IL-2, IL-6, IL-7, IL-8, IL-10, IL-15, TNF alpha, and granulocyte-macrophage colony-stimulating factor (GM-CSF).
Time Frame: Baseline up to Month 3
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 2 (Safety Management Study): Cohort 4 | Phase 2 (Safety Management Study): Cohort 5 | Phase 2 (Safety Management Study): Cohort 6
Number analyzed (Participants) | 41 | 50 | 40
pg/mL
  IP-10 | 1549.70 [469.20 to 2000.00] | 1746.15 [349.80 to 2000.00] | 1560.03 [347.00 to 2000.000]
  Granzyme B | 23.10 [1.00 to 322.60] | 27.90 [1.00 to 375.76] | 18.40 [1.00 to 162.30]
  IFN-gamma | 334.50 [24.90 to 1876.00] | 314.90 [7.50 to 1876.00] | 207.95 [18.80 to 1876.00]
  IL-1 RA: number analyzed (Participants) | 31 | 50 | 40
  IL-1 RA | 1093.70 [193.30 to 4493.10] | 908.00 [229.00 to 9000.00] | 1279.50 [227.00 to 9000.00]
  IL-2 | 11.20 [0.90 to 79.40] | 11.85 [0.90 to 142.70] | 8.40 [0.90 to 277.60]
  IL-6 | 136.70 [1.60 to 976.00] | 97.95 [1.60 to 976.00] | 47.25 [1.60 to 976.00]
  IL-7 | 33.10 [18.00 to 67.50] | 29.80 [1.40 to 65.20] | 28.25 [13.20 to 74.30]
  IL-8 | 67.40 [8.50 to 750.00] | 75.10 [5.80 to 750.00] | 52.55 [10.00 to 750.00]
  IL-10 | 19.60 [1.40 to 466.00] | 14.45 [0.70 to 300.90] | 13.30 [0.70 to 171.20]
  IL-15 | 45.80 [22.30 to 272.70] | 34.15 [1.40 to 140.00] | 37.20 [9.50 to 86.30]
  TNF alpha | 5.70 [2.00 to 54.60] | 5.25 [1.40 to 33.30] | 4.80 [2.10 to 20.20]
  GM-CSF | 4.40 [1.90 to 47.00] | 2.90 [1.90 to 35.60] | 1.90 [1.90 to 47.40]

22. Secondary Outcome: Pharmacodynamics: Peak Level of Cytokines (Ferritin, ICAM-1, IL-2 R, Perforin, and VCAM-1) in Serum (Phase 2 Cohorts 4, 5, and 6)
Description: Peak was defined as the maximum post-baseline level of the cytokine. Following key cytokines were measured: Ferritin, ICAM-1, IL-2 R, Perforin, and VCAM-1.
Time Frame: Baseline up to Month 3
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Phase 2 (Safety Management Study): Cohort 4 | Phase 2 (Safety Management Study): Cohort 5 | Phase 2 (Safety Management Study): Cohort 6
Number analyzed (Participants) | 41 | 50 | 40
ng/mL
  Ferritin | 1086.36 [95.55 to 23900] | 1516.11 [89.29 to 31600] | 903.50 [171.61 to 6555.10]
  ICAM-1 | 907.97 [359.51 to 5141.64] | 636.74 [361.38 to 4835.93] | 654.81 [355.15 to 4419.09]
  IL-2 R | 10.78 [2.81 to 94.59] | 7.82 [1.36 to 83.60] | 6.43 [1.70 to 33.31]
  Perforin | 17.22 [3.88 to 44.42] | 10.85 [2.53 to 100.00] | 10.12 [1.97 to 39.62]
  VCAM-1 | 1255.32 [594.51 to 3932.61] | 854.63 [476.60 to 6501.14] | 836.04 [411.93 to 5079.25]

23. Secondary Outcome: Pharmacodynamics: Peak Level of Cytokine (CRP) in Serum
Description: Peak was defined as the maximum post-baseline level of the cytokine.
Time Frame: Baseline up to Month 3
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Full Range); unit: mg/mL
Arm/Group | Phase 1 Study: Axicabtagene Ciloleucel and Conditioning Chemotherapy | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2 | Phase 2 (Safety Management Study): Cohort 3 | Phase 2 (Safety Management Study): Cohort 4 | Phase 2 (Safety Management Study): Cohort 5 | Phase 2 (Safety Management Study): Cohort 6
Number analyzed (Participants) | 7 | 77 | 24 | 38 | 41 | 50 | 40
mg/mL | 112.6 [14.6 to 655.0] | 215.7 [31.0 to 496.0] | 186.6 [18.5 to 496.0] | 137.8 [2.1 to 496.0] | 126.53 [18.19 to 496.00] | 74.84 [1.81 to 496.00] | 76.11 [7.31 to 496.00]

24. Secondary Outcome: Pharmacodynamics: Peak Level of Cytokine (Ferritin) in Serum (Phase 1 and Phase 2 Cohorts 1 and 2)
Description: Peak was defined as the maximum post-baseline level of the cytokine.
Time Frame: Baseline up to Month 3
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 1 Study: Axicabtagene Ciloleucel and Conditioning Chemotherapy | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2
Number analyzed (Participants) | 7 | 77 | 24
pg/mL | 1973400.0 [1201900.0 to 32984400.0] | 3681400.0 [780.0 to 25000000.0] | 1979360.0 [780.0 to 25000000.0]

25. Secondary Outcome: Pharmacodynamics: Peak Level of Cytokine (Ferritin) in Serum (Phase 2 Cohort 3)
Description: Peak was defined as the maximum post-baseline level of the cytokine.
Time Frame: Baseline up to Month 3
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Phase 2 (Safety Management Study): Cohort 3
Number analyzed (Participants) | 38
ng/mL | 2440.2 [0.8 to 25000.0]

26. Secondary Outcome: Percentage of Participants With Positive Replication Competent Retrovirus (RCR)
Description: RCR was analyzed in blood samples by central laboratory. Because axicabtagene ciloleucel comprised retroviral vector transduced T cells, the presence of RCR in the blood of treated participants was reported.
Time Frame: Day 0 (pre-infusion) up to last follow-up visit (maximum duration: 7.7, 6.8, 5.4, 4.4, 4.1 years for Phase 1 and Phase 2 Cohorts 1, 2, 3, 4, 5, and 6 respectively)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 Study: Axicabtagene Ciloleucel and Conditioning Chemotherapy | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2 | Phase 2 (Safety Management Study): Cohort 3 | Phase 2 (Safety Management Study): Cohort 4 | Phase 2 (Safety Management Study): Cohort 5 | Phase 2 (Safety Management Study): Cohort 6
Number analyzed (Participants) | 7 | 77 | 24 | 38 | 41 | 50 | 40
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Phase 2 Safety Management Study: Number of Participants With the European Quality of Life Five Dimension Five Level Scale (EQ-5D) Score
Description: EQ-5D is a self-reported questionnaire used for assessing the overall health status of a participant scoring 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension was divided into 5 levels of severity: "No problem", "Slight problems", "Moderate problems", "Severe problems", and "Extreme problems (unable to perform)". EQ-5D health states, defined by the EQ-5D descriptive system, are converted into a single summary index by applying a formula that attaches values (also called QOL weights or QOL utilities) to each of the levels in each dimension. EQ-5D Summary Index values range from -0.11 (worst health state) to 1.00 (perfect health state).
Time Frame: Baseline, Week 4, Month 3, and Month 6
Population: Participants in Safety Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 (Safety Management Study): Cohort 3 | Phase 2 (Safety Management Study): Cohort 4 | Phase 2 (Safety Management Study): Cohort 5 | Phase 2 (Safety Management Study): Cohort 6
Number analyzed (Participants) | 38 | 39 | 47 | 34
Participants
  Baseline: Mobility: No problem | 30 | 25 | 33 | 26
  Baseline: Mobility: Slight problem | 7 | 9 | 5 | 4
  Baseline: Mobility: Moderate problem | 1 | 5 | 7 | 3
  Baseline: Mobility: Severe problem | 0 | 0 | 1 | 1
  Baseline: Mobility: Unable to perform | 0 | 0 | 1 | 0
  Week 4: Mobility: number analyzed (Participants) | 32 | 37 | 38 | 29
  Week 4: Mobility: No problem | 16 | 21 | 23 | 20
  Week 4: Mobility: Slight problem | 11 | 7 | 9 | 5
  Week 4: Mobility: Moderate problem | 4 | 5 | 4 | 4
  Week 4: Mobility: Severe problem | 0 | 3 | 1 | 0
  Week 4: Mobility: Unable to perform | 1 | 1 | 1 | 0
  Month 3: Mobility: number analyzed (Participants) | 23 | 31 | 33 | 29
  Month 3: Mobility: No problem | 14 | 20 | 21 | 22
  Month 3: Mobility: Slight problem | 6 | 8 | 6 | 3
  Month 3: Mobility: Moderate problem | 2 | 2 | 6 | 3
  Month 3: Mobility: Severe problem | 1 | 1 | 0 | 1
  Month 3: Mobility: Unable to perform | 0 | 0 | 0 | 0
  Month 6: Mobility: number analyzed (Participants) | 18 | 25 | 17 | 27
  Month 6: Mobility: No problem | 10 | 19 | 11 | 15
  Month 6: Mobility: Slight problem | 6 | 4 | 2 | 8
  Month 6: Mobility: Moderate problem | 2 | 2 | 4 | 3
  Month 6: Mobility: Severe problem | 0 | 0 | 0 | 1
  Month 6: Mobility: Unable to perform | 0 | 0 | 0 | 0
  Baseline: Self-care: No problem | 37 | 38 | 44 | 32
  Baseline: Self-care: Slight problem | 1 | 1 | 3 | 1
  Baseline: Self-care: Moderate problem | 0 | 0 | 0 | 1
  Baseline: Self-care: Severe problem | 0 | 0 | 0 | 0
  Baseline: Self-care: Unable to perform | 0 | 0 | 0 | 0
  Week 4: Self-care: number analyzed (Participants) | 32 | 37 | 38 | 29
  Week 4: Self-care: No problem | 25 | 33 | 31 | 24
  Week 4: Self-care: Slight problem | 5 | 3 | 6 | 3
  Week 4: Self-care: Moderate problem | 1 | 0 | 1 | 1
  Week 4: Self-care: Severe problem | 0 | 1 | 0 | 1
  Week 4: Self-care: Unable to perform | 1 | 0 | 0 | 0
  Month 3: Self-care: number analyzed (Participants) | 23 | 31 | 33 | 29
  Month 3: Self-care: No problem | 19 | 29 | 32 | 25
  Month 3: Self-care: Slight problem | 4 | 2 | 1 | 4
  Month 3: Self-care: Moderate problem | 0 | 0 | 0 | 0
  Month 3: Self-care: Severe problem | 0 | 0 | 0 | 0
  Month 3: Self-care: Unable to perform | 0 | 0 | 0 | 0
  Month 6: Self-care: number analyzed (Participants) | 18 | 25 | 17 | 27
  Month 6: Self-care: No problem | 17 | 25 | 16 | 20
  Month 6: Self-care: Slight problem | 1 | 0 | 1 | 7
  Month 6: Self-care: Moderate problem | 0 | 0 | 0 | 0
  Month 6: Self-care: Severe problem | 0 | 0 | 0 | 0
  Month 6: Self-care: Unable to perform | 0 | 0 | 0 | 0
  Baseline: Usual activities: No problem | 22 | 22 | 24 | 16
  Baseline: Usual activities: Slight problem | 10 | 6 | 13 | 14
  Baseline: Usual activities: Moderate problem | 4 | 8 | 8 | 2
  Baseline: Usual activities: Severe problem | 2 | 1 | 1 | 2
  Baseline: Usual activities: Unable to perform | 0 | 2 | 1 | 0
  Week 4: Usual activities: number analyzed (Participants) | 32 | 37 | 37 | 29
  Week 4: Usual activities: No problem | 6 | 12 | 12 | 12
  Week 4: Usual activities: Slight problem | 13 | 11 | 13 | 11
  Week 4: Usual activities: Moderate problem | 11 | 8 | 8 | 4
  Week 4: Usual activities: Severe problem | 0 | 3 | 2 | 1
  Week 4: Usual activities: Unable to perform | 2 | 3 | 2 | 1
  Month 3: Usual activities: number analyzed (Participants) | 23 | 31 | 33 | 29
  Month 3: Usual activities: No problem | 8 | 16 | 19 | 12
  Month 3: Usual activities: Slight problem | 9 | 9 | 10 | 14
  Month 3: Usual activities: Moderate problem | 5 | 5 | 2 | 2
  Month 3: Usual activities: Severe problem | 1 | 1 | 1 | 1
  Month 3: Usual activities: Unable to perform | 0 | 0 | 1 | 0
  Month 6: Usual activities: number analyzed (Participants) | 18 | 25 | 17 | 27
  Month 6: Usual activities: No problem | 9 | 15 | 10 | 11
  Month 6: Usual activities: Slight problem | 5 | 7 | 4 | 12
  Month 6: Usual activities: Moderate problem | 3 | 3 | 2 | 3
  Month 6: Usual activities: Severe problem | 1 | 0 | 1 | 0
  Month 6: Usual activities: Unable to perform | 0 | 0 | 0 | 1
  Baseline: Pain/Discomfort: No problem | 18 | 17 | 16 | 15
  Baseline: Pain/Discomfort: Slight problem | 9 | 17 | 18 | 14
  Baseline: Pain/Discomfort: Moderate problem | 8 | 5 | 7 | 4
  Baseline: Pain/Discomfort: Severe problem | 1 | 0 | 5 | 1
  Baseline: Pain/Discomfort: Unable to perform | 2 | 0 | 1 | 0
  Week 4: Pain/Discomfort: number analyzed (Participants) | 32 | 37 | 37 | 29
  Week 4: Pain/Discomfort: No problem | 12 | 19 | 20 | 17
  Week 4: Pain/Discomfort: Slight problem | 12 | 13 | 10 | 9
  Week 4: Pain/Discomfort: Moderate problem | 7 | 2 | 5 | 3
  Week 4: Pain/Discomfort: Severe problem | 1 | 3 | 2 | 0
  Week 4: Pain/Discomfort: Unable to perform | 0 | 0 | 0 | 0
  Month 3: Pain/Discomfort: number analyzed (Participants) | 23 | 31 | 33 | 29
  Month 3: Pain/Discomfort: No problem | 9 | 10 | 18 | 16
  Month 3: Pain/Discomfort: Slight problem | 5 | 14 | 9 | 5
  Month 3: Pain/Discomfort: Moderate problem | 9 | 6 | 6 | 5
  Month 3: Pain/Discomfort: Severe problem | 0 | 1 | 0 | 3
  Month 3: Pain/Discomfort: Unable to perform | 0 | 0 | 0 | 0
  Month 6: Pain/Discomfort: number analyzed (Participants) | 17 | 25 | 17 | 27
  Month 6: Pain/Discomfort: No problem | 8 | 9 | 6 | 12
  Month 6: Pain/Discomfort: Slight problem | 4 | 14 | 8 | 8
  Month 6: Pain/Discomfort: Moderate problem | 5 | 1 | 3 | 4
  Month 6: Pain/Discomfort: Severe problem | 0 | 1 | 0 | 3
  Month 6: Pain/Discomfort: Unable to perform | 0 | 0 | 0 | 0
  Baseline: Anxiety/Depression: No problem | 16 | 23 | 18 | 21
  Baseline: Anxiety/Depression: Slight problem | 16 | 13 | 17 | 9
  Baseline: Anxiety/Depression: Moderate problem | 3 | 3 | 10 | 3
  Baseline: Anxiety/Depression: Severe problem | 1 | 0 | 1 | 1
  Baseline: Anxiety/Depression: Unable to perform | 2 | 0 | 1 | 0
  Week 4: Anxiety/Depression: number analyzed (Participants) | 32 | 37 | 38 | 29
  Week 4: Anxiety/Depression: No problem | 9 | 25 | 21 | 23
  Week 4: Anxiety/Depression: Slight problem | 15 | 8 | 12 | 3
  Week 4: Anxiety/Depression: Moderate problem | 7 | 3 | 5 | 3
  Week 4: Anxiety/Depression: Severe problem | 1 | 1 | 0 | 0
  Week 4: Anxiety/Depression: Unable to perform | 0 | 0 | 0 | 0
  Month 3: Anxiety/Depression: number analyzed (Participants) | 23 | 31 | 33 | 29
  Month 3: Anxiety/Depression: No problem | 11 | 19 | 16 | 19
  Month 3: Anxiety/Depression: Slight problem | 5 | 8 | 12 | 7
  Month 3: Anxiety/Depression: Moderate problem | 6 | 4 | 4 | 2
  Month 3: Anxiety/Depression: Severe problem | 1 | 0 | 1 | 1
  Month 3: Anxiety/Depression: Unable to perform | 0 | 0 | 0 | 0
  Month 6: Anxiety/Depression: number analyzed (Participants) | 18 | 25 | 17 | 26
  Month 6: Anxiety/Depression: No problem | 9 | 14 | 7 | 18
  Month 6: Anxiety/Depression: Slight problem | 5 | 10 | 8 | 5
  Month 6: Anxiety/Depression: Moderate problem | 3 | 0 | 1 | 3
  Month 6: Anxiety/Depression: Severe problem | 0 | 1 | 1 | 0
  Month 6: Anxiety/Depression: Unable to perform | 1 | 0 | 0 | 0

28. Secondary Outcome: Phase 2 Safety Management Study: EQ-5D Visual Analogue Scale (VAS) Score
Description: EQ-5D is a self-reported questionnaire used for assessing the overall health status of a participant. The EQ-5D-VAS records the participant's self-rated health on a vertical visual analogue scale and is asked to make a global assessment of their current state of health with 0 indicating the worst health they can imagine and 100 indicating the best health they can imagine.
Time Frame: Baseline, Week 4, Month 3, and Month 6
Population: Participants in Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 2 (Safety Management Study): Cohort 3 | Phase 2 (Safety Management Study): Cohort 4 | Phase 2 (Safety Management Study): Cohort 5 | Phase 2 (Safety Management Study): Cohort 6
Number analyzed (Participants) | 38 | 38 | 47 | 34
units on a scale
  Baseline | 71.2 (21.3) | 69.5 (18.8) | 66.7 (20.7) | 70.9 (17.0)
  Week 4: number analyzed (Participants) | 32 | 36 | 38 | 29
  Week 4 | 67.8 (15.6) | 67.2 (20.9) | 70.8 (14.8) | 76.1 (13.2)
  Month 3: number analyzed (Participants) | 23 | 31 | 33 | 29
  Month 3 | 74.9 (16.6) | 78.8 (14.7) | 73.3 (19.9) | 76.5 (15.0)
  Month 6: number analyzed (Participants) | 18 | 25 | 17 | 27
  Month 6 | 77.1 (21.4) | 85.1 (12.1) | 77.1 (14.7) | 79.8 (14.0)

ADVERSE EVENTS:
Time Frame: Adverse event: Up to 7.7 years; All-cause mortality: Enrollment up to last follow up visit (maximum duration: 7.7 years; The number of deaths reported in the Participant Flow for Phase 2 Cohort 1 (53) is more than the number of deaths reported in the All-Cause Mortality for Phase 2 Cohort 1 (49) within the table below because the deaths that occurred in the main phase and retreatment phase arms are being reported separately.
Description: Adverse events: For Phase 1 and Phase 2 (Cohorts 1 to 6): The Safety Analysis Set included all participants treated with any dose of axicabtagene ciloleucel; For retreatment groups: The Safety-Retreatment Analysis Set include all participants with re-treatment of axicabtagene ciloleucel. All-cause mortality: For Phase 1 and Phase 2 (Cohorts 1 to 6): All Enrolled Analysis Set included all enrolled participants; Retreatment groups,participants were included from Safety-Retreatment Analysis Set.
Groups:
- Retreatment Axicabtagene Ciloleucel: Phase 1: Participants who initially responded and subsequently relapsed, became eligible for second course of conditioning chemotherapy and axicabtagene ciloleucel. Participants received the axicabtagene ciloleucel regimen selected for Phase 2.
- Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 1; Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 2; Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 3; Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 4; Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 5; Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 6: Participants who initially responded and subsequently relapsed, became eligible for second course of conditioning chemotherapy and axicabtagene ciloleucel. Participants received the same axicabtagene ciloleucel regimen as the original target dose.
Arm/Group | Phase 1 Study: Axicabtagene Ciloleucel and Conditioning Chemotherapy | Phase 2 (Pivotal Study): Cohort 1 | Phase 2 (Pivotal Study): Cohort 2 | Phase 2 (Safety Management Study): Cohort 3 | Phase 2 (Safety Management Study): Cohort 4 | Phase 2 (Safety Management Study): Cohort 5 | Phase 2 (Safety Management Study): Cohort 6 | Retreatment Axicabtagene Ciloleucel: Phase 1 | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 1 | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 2 | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 3 | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 4 | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 5 | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 6
All-Cause Mortality (participants affected / at risk) | 5/8 | 49/81 | 13/30 | 23/42 | 20/46 | 37/58 | 20/42 | 1/1 | 8/9 | 2/2 | 1/2 | 2/2 | 2/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 5/7 | 40/77 | 14/24 | 26/38 | 24/41 | 27/50 | 25/40 | 1/1 | 5/9 | 1/2 | 2/2 | 0/2 | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 7/7 | 77/77 | 23/24 | 38/38 | 41/41 | 50/50 | 40/40 | 1/1 | 9/9 | 2/2 | 2/2 | 2/2 | 2/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Study: Axicabtagene Ciloleucel and Conditioning Chemotherapy (N=7) | Phase 2 (Pivotal Study): Cohort 1 (N=77) | Phase 2 (Pivotal Study): Cohort 2 (N=24) | Phase 2 (Safety Management Study): Cohort 3 (N=38) | Phase 2 (Safety Management Study): Cohort 4 (N=41) | Phase 2 (Safety Management Study): Cohort 5 (N=50) | Phase 2 (Safety Management Study): Cohort 6 (N=40) | Retreatment Axicabtagene Ciloleucel: Phase 1 (N=1) | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 1 (N=9) | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 2 (N=2) | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 3 (N=2) | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 4 (N=2) | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 5 (N=2) | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 6 (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 5 | 1 | 3 | 2 | 5 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus enteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Human herpesvirus 6 encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 7 | 3 | 1 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotavirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin T increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amyotrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 0 | 3 | 3 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 3 | 1 | 1 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Apraxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgraphia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspraxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 16 | 3 | 9 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine with aura (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Quadriplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure like phenomena (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 3 | 0 | 2 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 3 | 2 | 3 | 1 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Reexpansion pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 1 | 4 | 2 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Study: Axicabtagene Ciloleucel and Conditioning Chemotherapy (N=7) | Phase 2 (Pivotal Study): Cohort 1 (N=77) | Phase 2 (Pivotal Study): Cohort 2 (N=24) | Phase 2 (Safety Management Study): Cohort 3 (N=38) | Phase 2 (Safety Management Study): Cohort 4 (N=41) | Phase 2 (Safety Management Study): Cohort 5 (N=50) | Phase 2 (Safety Management Study): Cohort 6 (N=40) | Retreatment Axicabtagene Ciloleucel: Phase 1 (N=1) | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 1 (N=9) | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 2 (N=2) | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 3 (N=2) | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 4 (N=2) | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 5 (N=2) | Retreatment Axicabtagene Ciloleucel: Phase 2 Cohort 6 (N=0)
Anaemia (Blood and lymphatic system disorders) | 4 | 47 | 13 | 22 | 19 | 19 | 13 | 1 | 3 | 1 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 21 | 8 | 10 | 3 | 2 | 2 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 13 | 3 | 4 | 7 | 8 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 5 | 0 | 0 | 3 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 26 | 12 | 18 | 16 | 16 | 20 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 24 | 6 | 12 | 7 | 9 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 5 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 5 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 19 | 2 | 4 | 2 | 3 | 5 | 0 | 4 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 3 | 29 | 8 | 6 | 7 | 7 | 6 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid function disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 2 | 2 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 5 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 8 | 3 | 3 | 2 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 15 | 5 | 7 | 6 | 8 | 15 | 1 | 3 | 2 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 29 | 8 | 16 | 25 | 11 | 11 | 0 | 2 | 2 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 7 | 3 | 3 | 2 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 4 | 0 | 5 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 22 | 12 | 15 | 12 | 12 | 14 | 1 | 4 | 0 | 1 | 2 | 2 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 17 | 11 | 9 | 6 | 7 | 8 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Asthenia (General disorders) | 0 | 5 | 2 | 3 | 2 | 4 | 5 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 32 | 7 | 11 | 11 | 14 | 8 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 34 | 12 | 18 | 19 | 12 | 18 | 0 | 3 | 0 | 1 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 2 | 0 | 4 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 4 | 0 | 1 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 5 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 12 | 2 | 6 | 2 | 3 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 5 | 1 | 5 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 7 | 66 | 21 | 35 | 39 | 40 | 33 | 1 | 9 | 2 | 1 | 2 | 2 | 0
Swelling (General disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 3 | 10 | 3 | 2 | 6 | 1 | 8 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 1 | 4 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 3 | 3 | 1 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 4 | 0 | 1 | 6 | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 3 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 5 | 4 | 7 | 3 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 3 | 1 | 0 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 5 | 2 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 13 | 5 | 8 | 5 | 7 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 11 | 5 | 7 | 4 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 3 | 1 | 4 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 3 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 4 | 2 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood immunoglobulin G decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 2 | 5 | 7 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immunoglobulins decreased (Investigations) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 12 | 6 | 4 | 4 | 8 | 7 | 1 | 3 | 2 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 27 | 7 | 11 | 13 | 25 | 14 | 0 | 4 | 2 | 0 | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 2 | 25 | 5 | 9 | 10 | 17 | 6 | 1 | 3 | 1 | 0 | 1 | 1 | 0
Serum ferritin increased (Investigations) | 0 | 1 | 1 | 2 | 3 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 11 | 4 | 1 | 0 | 4 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 4 | 0 | 1 | 4 | 4 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 2 | 23 | 8 | 10 | 6 | 14 | 10 | 1 | 3 | 2 | 0 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 31 | 12 | 10 | 3 | 6 | 8 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 5 | 4 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 12 | 6 | 2 | 1 | 0 | 4 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 6 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 22 | 9 | 4 | 2 | 0 | 2 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 23 | 11 | 4 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 23 | 8 | 6 | 6 | 10 | 11 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 5 | 4 | 6 | 2 | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 20 | 10 | 2 | 2 | 1 | 6 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 19 | 6 | 5 | 6 | 5 | 11 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 12 | 2 | 1 | 4 | 4 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 13 | 2 | 1 | 5 | 4 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 1 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 11 | 2 | 4 | 1 | 2 | 6 | 0 | 3 | 1 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 10 | 3 | 5 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 7 | 4 | 1 | 4 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 13 | 4 | 8 | 4 | 9 | 4 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Apraxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 12 | 9 | 5 | 7 | 8 | 6 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 3 | 1 | 3 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dysgraphia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 4 | 20 | 6 | 9 | 5 | 5 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 34 | 12 | 19 | 16 | 17 | 13 | 0 | 3 | 1 | 0 | 2 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 6 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 4 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Poor sucking reflex (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 3 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 3 | 10 | 4 | 3 | 5 | 5 | 5 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 4 | 23 | 6 | 16 | 5 | 11 | 9 | 0 | 4 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 5 | 3 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 9 | 3 | 4 | 0 | 2 | 4 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 19 | 8 | 16 | 4 | 6 | 12 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 1 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 4 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 7 | 2 | 4 | 2 | 0 | 6 | 1 | 3 | 1 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 4 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 6 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 2 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 4 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 0 | 2 | 2 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 7 | 1 | 4 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 4 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 18 | 6 | 9 | 11 | 6 | 6 | 0 | 5 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 11 | 4 | 5 | 3 | 4 | 8 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 24 | 5 | 9 | 6 | 5 | 7 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 2 | 1 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2 | 2 | 1 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 9 | 1 | 5 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 6 | 2 | 1 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 2 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Capillary leak syndrome (Vascular disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 9 | 4 | 2 | 2 | 3 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 3 | 44 | 14 | 22 | 24 | 25 | 21 | 1 | 1 | 1 | 0 | 1 | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol: Amendment 8 (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT02348216/Prot_000.pdf
  • Study Protocol: Amendment 10 (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT02348216/Prot_002.pdf
  • Statistical Analysis Plan (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT02348216/SAP_001.pdf